CLINICAL TRIAL: NCT00705432
Title: A Phase 3, Safety and Efficacy Study of Boceprevir in Previously Untreated Subjects With Chronic Hepatitis C Genotype 1
Brief Title: Safety and Efficacy of Boceprevir in Previously Untreated Subjects With Chronic Hepatitis C Genotype 1 (Study P05216AM2) (COMPLETED)
Acronym: SPRINT-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05216; EUDRACT # 2007-005508-42; NCT00795431 (obsolete NCT alias)
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. Placebo + PEG + RBV (Placebo Comparator): PegIntron (PEG) 1.5 μg/kg + Ribavirin (RBV) (weight-based dosing [WBD]) for 4 weeks (lead in treatment) followed by placebo + PEG 1.5 μg/kg + RBV (WBD) for 44 weeks with 24 weeks post-treatment follow-up.
  Interventions: Biological: Peginterferon alfa-2b (PEG); Drug: Ribavirin (RBV); Drug: Placebo
- 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) (Experimental): PEG 1.5 μg/kg + RBV (WBD) for 4 weeks (lead in treatment) followed by boceprevir + PEG 1.5 μg/kg + RBV (WBD) for 24 weeks. Participants were offered a response guided therapy (RGT) at treatment week 28.
  * At the Treatment Week 28 visit, participants whose HCV-RNA was undetectable from Treatment Weeks 8 to Treatment Week 24, will proceed to the 44-week follow-up.
  * At the Treatment Week 28 visit, participants with detectable HCV-RNA at Treatment Week 8 or at any subsequent assays will continue on therapy with placebo + PEG 1.5 μg/kg + RBV (WBD) for an additional 20 weeks, to complete a total of 48 weeks on treatment with 24 weeks post-treatment follow-up.
  Interventions: Biological: Peginterferon alfa-2b (PEG); Drug: Ribavirin (RBV); Drug: Boceprevir
- 3. Boceprevir + PEG + RBV - 44 Weeks (Experimental): PEG 1.5 μg/kg + RBV (WBD) for 4 weeks (lead in treatment) followed by boceprevir + PEG 1.5 μg/kg + RBV (WBD) for 44 weeks with 24 weeks post-treatment follow-up.
  Interventions: Biological: Peginterferon alfa-2b (PEG); Drug: Ribavirin (RBV); Drug: Boceprevir

INTERVENTIONS:
Biological: Peginterferon alfa-2b (PEG) — Peginterferon alfa-2b 1.5 μg/kg/week subcutaneously (SC)
  Other Names: PegIntron; PEG; SCH 54031
Drug: Ribavirin (RBV) — Ribavirin weight-based dosing (WBD) 600 mg/day to 1400 mg/day administered orally, divided twice daily (BID).
  Other Names: Rebetol; RBV; SCH 18908
Drug: Placebo — Placebo to boceprevir, 800 mg (4 x 200mg capsules) administered orally three times a day (TID).
  Arms: 1. Placebo + PEG + RBV
Drug: Boceprevir — Boceprevir, 800 mg (4 x 200 mg capsules) administered orally TID.
  Other Names: SCH 503034, Victrelis
  Arms: 2. Boceprevir + PEG + RBV - 24 Weeks (RGT); 3. Boceprevir + PEG + RBV - 44 Weeks

SUMMARY:
This study involves treatment with boceprevir or placebo in combination with PegIntron (PEG) + Ribavirin (RBV) (weight-based dosing [WBD]) in previously untreated adult participants with chronic hepatitis C (CHC) genotype 1. It is hypothesized that the addition of a third active anti- Hepatitis C Virus (anti-HCV) drug may lead to more rapid viral response than therapy with two drugs, and therefore, the addition of boceprevir to PegIntron plus ribavirin therapy after a 4-week lead-in period may allow for both increased rates of sustained virologic response (SVR) and shorter treatment durations (in some populations) than treatment with PegIntron plus ribavirin alone.

The study includes two separate cohorts, Cohort I (White participants) and Cohort II (Black participants). Participants from each cohort are assigned (randomized) to one of three study arms, all of which have a 4-week lead-in period with (PEG + RBV).

DETAILED DESCRIPTION:
Participants from Cohort I and Cohort II are assigned (randomized) to one of three study arms, all of which have a 4-week lead-in period with (PEG + RBV).

1. Control arm, participants are treated with (PEG + RBV + placebo) for 44 weeks after the lead-in.
2. Experimental arm with Response Guided Therapy (RGT)

   In this experimental arm, participants are treated with all three drugs (PEG + RBV + boceprevir) for 24 weeks after the lead-in. At treatment week 28, those participants with undetectable Hepatitis C Virus - ribonucleic acid (HCV-RNA) from week 8 (up to treatment week 24), will be considered to complete treatment, and will enter follow-up. Participants with detectable for HCV-RNA at week 8 or later will receive an additional 20 weeks of therapy with PegIntron and Ribavirin (PEG + RBV + placebo).
3. Experimental arm, participants are treated with all three drugs (PEG + RBV + Ribavirin) for 44 weeks after the lead-in.

All participants were followed up to 72 weeks following randomization.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have previously documented CHC genotype 1 infection.
* Participant must have a liver biopsy with histology consistent with CHC and no other etiology.
* Participants with bridging fibrosis or cirrhosis must have an ultrasound within 6 months of the Screening Visit (or between Screening and Day 1) with no findings suspicious for hepatocellular carcinoma (HCC).
* Participant must be >=18 years of age.
* Participant must weigh between 40 kg and 125 kg.
* Participant and participant's partner(s) must each agree to use acceptable methods of contraception for at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study drug, or longer if dictated by local regulations.
* Participants must be willing to give written informed consent.

Exclusion Criteria:

* Coinfection with the human immunodeficiency virus (HIV) or hepatitis B virus (HBsAg positive).
* Participants who received prior treatment for hepatitis C; other than herbal remedies, except those with known hepatotoxicity.
* Treatment with any investigational drug within 30 days of the randomization visit in this study.
* Participation in any other clinical trial within 30 days of randomization or intention to participate in another clinical trial during participation in this study.
* Evidence of decompensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy.
* Diabetic and/or hypertensive participants with clinically significant ocular examination findings: retinopathy, cotton wool spots, optic nerve disorder, retinal hemorrhage, or any other clinically significant abnormality.
* Pre-existing psychiatric condition(s).
* Clinical diagnosis of substance abuse of the specified drugs within the specified timeframes.
* Any known pre-existing medical condition that could interfere with the participant's participation in and completion of the study.
* Evidence of active or suspected malignancy, or a history of malignancy, within the last 5 years (except adequately treated carcinoma in situ and basal cell carcinoma of the skin). Participants under evaluation for malignancy are not eligible.
* Participants who are pregnant or nursing. Participants who intend to become pregnant during the study period. Male participants with partners who are, or intend to become, pregnant during the study period.
* Any other condition which, in the opinion of a physician, would make the participant unsuitable for enrollment or could interfere with the participant participating in and completing the study.
* Participants who are part of the site personnel directly involved with this study.
* Participants who are family members of the investigational study staff.
* Participants who had life-threatening serious adverse event (SAE) during screening period.
* Protocol-specified hematologic, biochemical, and serologic criteria: Hemoglobin <12 g/dL for females and <13 g/dL for males; Neutrophils <1500/mm^3 (blacks: <1200/mm^3); Platelets <100,000/mm^3; Direct bilirubin >1.5 x upper limit of normal (ULN)
* Serum albumin < lower limit of normal (LLN)
* Thyroid-stimulating hormone (TSH) >1.2 x ULN or <0.8 x LLN of laboratory, with certain exceptions.
* Serum creatinine >ULN of the laboratory reference.
* Protocol-specified serum glucose concentrations.
* protocol-specified alpha fetoprotein levels.
* Prothrombin time/partial thromboplastin time (PT/PTT) values >10% above laboratory reference range.
* Anti-nuclear antibodies (ANA) >1:320.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1472 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Ferrante SA, Chhatwal J, Brass CA, El Khoury AC, Poordad F, Bronowicki JP, Elbasha EH. Boceprevir for previously untreated patients with chronic hepatitis C Genotype 1 infection: a US-based cost-effectiveness modeling study. BMC Infect Dis. 2013 Apr 27;13:190. doi: 10.1186/1471-2334-13-190. PMID 23621902
- [Derived] Poordad F, Bronowicki JP, Gordon SC, Zeuzem S, Jacobson IM, Sulkowski MS, Poynard T, Morgan TR, Molony C, Pedicone LD, Sings HL, Burroughs MH, Sniukiene V, Boparai N, Goteti VS, Brass CA, Albrecht JK, Bacon BR; SPRINT-2 and RESPOND-2 Investigators. Factors that predict response of patients with hepatitis C virus infection to boceprevir. Gastroenterology. 2012 Sep;143(3):608-618.e5. doi: 10.1053/j.gastro.2012.05.011. Epub 2012 May 21. PMID 22626609
- [Derived] Poordad F, McCone J Jr, Bacon BR, Bruno S, Manns MP, Sulkowski MS, Jacobson IM, Reddy KR, Goodman ZD, Boparai N, DiNubile MJ, Sniukiene V, Brass CA, Albrecht JK, Bronowicki JP; SPRINT-2 Investigators. Boceprevir for untreated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1195-206. doi: 10.1056/NEJMoa1010494. PMID 21449783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1472 participants were enrolled in this study.
Pre-assignment Details: 373 participants were screened but not randomized. 1099 participants were randomized. Only 1097 received at least one dose of PegIntron (PEG) + Ribavirin (RBV) (lead-in treatment).
Groups:
- Cohort I - 1. Placebo + PEG + RBV: Cohort I (White participants) treated with PegIntron (PEG) 1.5 μg/kg + Ribavirin (RBV) (weight-based dosing [WBD]) for 4 weeks followed by placebo + PEG 1.5 μg/kg + RBV (WBD) for 44 weeks with 24 weeks post-treatment follow-up.
- Cohort I - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT): Cohort I (White participants) treated with PEG 1.5 μg/kg + RBV (WBD) for 4 weeks followed by boceprevir + PEG 1.5 μg/kg + RBV (WBD) for 24 weeks. Participants were offered a response guided therapy (RGT) at treatment week 28.
  * At the Treatment Week 28 visit, participants whose HCV-RNA was undetectable at Treatment Week 8 and at all subsequent assays (up to Treatment Week 24), will proceed to the 44-week follow-up.
  * At the Treatment Week 28 visit, participants with detectable HCV-RNA at Treatment Week 8 or at any subsequent assays will continue on therapy with placebo + PEG 1.5 μg/kg + RBV (WBD) for an additional 20 weeks, to complete a total of 48 weeks on treatment with 24 weeks post-treatment follow-up.
- Cohort I - 3. Boceprevir + PEG + RBV - 44 Weeks: Cohort I (White participants) treated with PEG 1.5 μg/kg + RBV (WBD) for 4 weeks followed by boceprevir + PEG 1.5 μg/kg + RBV (WBD) for 44 weeks with 24 weeks post-treatment follow-up.
- Cohort II - 1. Placebo + PEG + RBV: Cohort II (Black participants) treated with PegIntron (PEG) 1.5 μg/kg + Ribavirin (RBV) (weight-based dosing [WBD]) for 4 weeks followed by placebo + PEG 1.5 μg/kg + RBV (WBD) for 44 weeks with 24 weeks post-treatment follow-up.
- Cohort II - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT): Cohort II (Black participants) treated with PEG 1.5 μg/kg + RBV (WBD) for 4 weeks followed by boceprevir + PEG 1.5 μg/kg + RBV (WBD) for 24 weeks. Participants were offered a response guided therapy (RGT) at treatment week 28.
  * At the Treatment Week 28 visit, participants whose HCV-RNA was undetectable at Treatment Week 8 and at all subsequent assays (up to Treatment Week 24), will proceed to the 44-week follow-up.
  * At the Treatment Week 28 visit, participants with detectable HCV-RNA at Treatment Week 8 or at any subsequent assays will continue on therapy with placebo + PEG 1.5 μg/kg + RBV (WBD) for an additional 20 weeks, to complete a total of 48 weeks on treatment with 24 weeks post-treatment follow-up.
- Cohort II - 3. Boceprevir + PEG + RBV - 44 Weeks: Cohort II (Black participants) treated with PEG 1.5 μg/kg + RBV (WBD) for 4 weeks followed by boceprevir + PEG 1.5 μg/kg + RBV (WBD) for 44 weeks with 24 weeks post-treatment follow-up.
Period: Treatment Period
Arm/Group | Cohort I - 1. Placebo + PEG + RBV | Cohort I - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort I - 3. Boceprevir + PEG + RBV - 44 Weeks | Cohort II - 1. Placebo + PEG + RBV | Cohort II - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort II - 3. Boceprevir + PEG + RBV - 44 Weeks
Started | 311 | 316 | 311 | 52 | 52 | 55
STARTED BOCEPREVIR/PLACEBO | 297 | 303 | 299 | 47 | 47 | 55
Completed | 148 | 205 | 190 | 11 | 24 | 25
Not Completed | 163 | 111 | 121 | 41 | 28 | 30
Not completed — Adverse Event | 45 | 37 | 51 | 12 | 8 | 9
Not completed — Treatment failure | 92 | 42 | 33 | 25 | 13 | 14
Not completed — Non medical reason | 26 | 32 | 37 | 4 | 7 | 7
Period: Follow-up Period (Upto Week 72)
Arm/Group | Cohort I - 1. Placebo + PEG + RBV | Cohort I - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort I - 3. Boceprevir + PEG + RBV - 44 Weeks | Cohort II - 1. Placebo + PEG + RBV | Cohort II - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort II - 3. Boceprevir + PEG + RBV - 44 Weeks
Started | 278 | 295 | 291 | 42 | 44 | 53
Completed | 207 | 252 | 266 | 28 | 38 | 46
Not Completed | 71 | 43 | 25 | 14 | 6 | 7
Not completed — Adverse Event | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Non medical reason | 69 | 42 | 24 | 14 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I - 1. Placebo + PEG + RBV | Cohort I - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort I - 3. Boceprevir + PEG + RBV - 44 Weeks | Cohort II - 1. Placebo + PEG + RBV | Cohort II - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort II - 3. Boceprevir + PEG + RBV - 44 Weeks | Total
Number analyzed (Participants) | 311 | 316 | 311 | 52 | 52 | 55 | 1097
Age, Customized [Number; unit: participants]
  <40 years | 51 | 45 | 49 | 6 | 3 | 4 | 158
  >= 40 and <65 years | 246 | 261 | 255 | 45 | 47 | 51 | 905
  >=65 years | 14 | 10 | 7 | 1 | 2 | 0 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 116 | 123 | 17 | 23 | 22 | 441
  Male | 171 | 200 | 188 | 35 | 29 | 33 | 656

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR) Rate
Description: Previously untreated adults with CHC genotype 1 were treated with the assigned study medication. Participants who had undetectable plasma HCV-RNA at FW 24 had achieved SVR. SVR rate is the percent of participants achieving SVR.
  HCV-RNA was detected by a nucleic acid amplification test and the limit of detection for this assay is 9.3 IU/mL.
  If a participant was missing data at FW 24 after having had undetectable HCV-RNA at FW 12, the participant was to be considered to have SVR.
Time Frame: At Follow-up Week (FW) 24
Population: Full analysis set (FAS). All randomized participants who received at least one dose of any study medication (PEG, RBV or boceprevir).
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort I - 1. Placebo + PEG + RBV | Cohort I - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort I - 3. Boceprevir + PEG + RBV - 44 Weeks | Cohort II - 1. Placebo + PEG + RBV | Cohort II - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort II - 3. Boceprevir + PEG + RBV - 44 Weeks
Number analyzed (Participants) | 311 | 316 | 311 | 52 | 52 | 55
Percentage of participants | 40.2 | 66.8 | 68.5 | 23.1 | 42.3 | 52.7
Statistical Analysis 1: Comparison: Cohort I - 1. Placebo + PEG + RBV vs Cohort I - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel Haenszel Chi-square test; Adjustments were made for for baseline stratification factors: viral load (>400,000 vs. ≤400,000 IU/mL) and Genotype (1a vs 1b); The difference in SVR = 26.6, 95% CI 2-sided [19.1 to 34.1]
Statistical Analysis 2: Comparison: Cohort I - 1. Placebo + PEG + RBV vs Cohort I - 3. Boceprevir + PEG + RBV - 44 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel Haenszel Chi-square test; Adjustments were made for baseline stratification factors: viral load (>400,000 vs. ≤400,000 IU/mL) and Genotype (1a vs 1b); The difference in SVR = 28.3, 95% CI 2-sided [20.8 to 35.8]
Statistical Analysis 3: Comparison: Cohort II - 1. Placebo + PEG + RBV vs Cohort II - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT); Test type: Superiority or Other; p = 0.0440, Cochran-Mantel Haenszel Chi-square test; Adjustments were made for the baseline stratification factors: viral load (>400,000 vs. ≤400,000 IU/mL) and Genotype (1a vs 1b); The difference in SVR = 19.2, 95% CI 2-sided [1.6 to 36.9]
Statistical Analysis 4: Comparison: Cohort II - 1. Placebo + PEG + RBV vs Cohort II - 3. Boceprevir + PEG + RBV - 44 Weeks; Test type: Superiority or Other; p = 0.0035, Cochran-Mantel Haenszel Chi-square; [statistical method as in outcome 1, analysis 3]; The difference in SVR = 29.7, 95% CI 2-sided [12.2 to 47.1]

2. Secondary Outcome: Sustained Virologic Response (SVR) Rate in Participants Treated With Study Drug (Boceprevir or Placebo)
Description: Previously untreated adults with CHC genotype 1 were treated with the assigned study medication. Participants who had undetectable plasma HCV-RNA at FW 24 had achieved SVR. SVR rate was the percentage of participants treated with at least one dose of boceprevir or placebo who had achieved SVR.
  HCV-RNA in participant's plasma samples was detected by a nucleic acid amplification assay with a limit of detection of 9.3 IU/mL.
  If a participant was missing data at FW 24 after having had undetectable HCV-RNA at FW 12, the participant was to be considered to have a SVR.
Time Frame: At FW 24
Population: Modified intent-to-treat set (mITT). All randomized participants who received at least one dose of boceprevir or placebo.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort I - 1. Placebo + PEG + RBV | Cohort I - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort I - 3. Boceprevir + PEG + RBV - 44 Weeks | Cohort II - 1. Placebo + PEG + RBV | Cohort II - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort II - 3. Boceprevir + PEG + RBV - 44 Weeks
Number analyzed (Participants) | 297 | 303 | 299 | 47 | 47 | 55
Percentage of participants | 42.1 | 69.6 | 71.2 | 25.5 | 46.8 | 52.7
Statistical Analysis 1: Comparison: Cohort I - 1. Placebo + PEG + RBV vs Cohort I - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel Haenszel Chi-square; [statistical method as in outcome 1, analysis 3]; The difference in SVR rates = 27.5, 95% CI 2-sided [19.2 to 35.2]
Statistical Analysis 2: Comparison: Cohort I - 1. Placebo + PEG + RBV vs Cohort I - 3. Boceprevir + PEG + RBV - 44 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel Haenszel Chi-square; [statistical method as in outcome 1, analysis 3]; The difference in SVR rates = 29.1, 95% CI 2-sided [21.5 to 36.8]
Statistical Analysis 3: Comparison: Cohort II - 1. Placebo + PEG + RBV vs Cohort II - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT); Test type: Superiority or Other; p = 0.0366, Cochran-Mantel Haenszel Chi-square test; [statistical method as in outcome 1, analysis 3]; The difference in SVR = 21.3, 95% CI 2-sided [2.3 to 40.2]
Statistical Analysis 4: Comparison: Cohort II - 1. Placebo + PEG + RBV vs Cohort II - 3. Boceprevir + PEG + RBV - 44 Weeks; Test type: Superiority or Other; p = 0.0107, Cochran-Mantel Haenszel Chi-square; [statistical method as in outcome 1, analysis 3]; The difference in SVR = 27.2, 95% CI 2-sided [9.0 to 45.3]

3. Secondary Outcome: Number of Participants With Undetectable HCV-RNA at Follow-up Week 12 and at 72 Weeks After Randomization.
Description: Previously untreated adults with CHC genotype 1 were treated with the assigned study medication. The number of participants who had undetectable plasma HCV-RNA at FW 12, and 72 weeks after randomization are reported.
  HCV-RNA was detected by a nucleic acid amplification test and the limit of detection for this assay is 9.3 IU/mL.
Time Frame: At FW 12 and at 72 weeks after randomization
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cohort I - 1. Placebo + PEG + RBV | Cohort I - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort I - 3. Boceprevir + PEG + RBV - 44 Weeks | Cohort II - 1. Placebo + PEG + RBV | Cohort II - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort II - 3. Boceprevir + PEG + RBV - 44 Weeks
Number analyzed (Participants) | 311 | 316 | 311 | 52 | 52 | 55
Participants
  At follow-up week 12 | 127 | 209 | 209 | 11 | 21 | 29
  72 weeks after randomization | 120 | 194 | 205 | 11 | 20 | 27

4. Secondary Outcome: Number of Participants With Early Virologic Response (Undetectable HCV-RNA at Treatment Week 2, 4, 8, 12, 16, or 20)
Description: Early virologic response was defined as undetectable HCV-RNA at in participants by treatment week 2, 4, 8, 12, 16, or 20.
  HCV-RNA in participant's plasma samples was detected by a nucleic acid amplification assay with a limit of detection of 9.3 IU/mL.
Time Frame: At Treatment Week 2, 4, 8, 12, 16, or 20
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cohort I - 1. Placebo + PEG + RBV | Cohort I - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort I - 3. Boceprevir + PEG + RBV - 44 Weeks | Cohort II - 1. Placebo + PEG + RBV | Cohort II - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort II - 3. Boceprevir + PEG + RBV - 44 Weeks
Number analyzed (Participants) | 311 | 316 | 311 | 52 | 52 | 55
Participants
  Treatment week 2 | 8 | 11 | 8 | 0 | 1 | 0
  Treatment week 4 | 28 | 18 | 20 | 2 | 1 | 0
  Treatment week 8 | 56 | 190 | 182 | 4 | 18 | 22
  Treatment week 12 | 108 | 237 | 231 | 10 | 25 | 33
  Treatment week 16 | 138 | 231 | 237 | 15 | 26 | 36
  Treatment week 20 | 157 | 231 | 231 | 15 | 27 | 32

5. Secondary Outcome: Number of Participants With Early Virologic Response (Undetectable HCV-RNA at Treatment Week 4, 8, 12, 16, or 20) Who Achieved SVR
Description: Participants with early virologic response were those who had undetectable HCV-RNA by treatment week 4, 8, 12, 16, or 20. Participants who had undetectable plasma HCV-RNA at FW 24 had SVR. The number of participants with early virologic response that also achieved SVR is reported.
  HCV-RNA in participant's plasma samples was detected by a nucleic acid amplification assay with a limit of detection of 9.3 IU/mL.
Time Frame: At Treatment Week 4, 8, 12, 16, 20
Population: Participants that had undetectable HCV RNA for the treatment weeks 4, 8, 12, 16, and 20.
Measure: Number; unit: Participants
Arm/Group | Cohort I - 1. Placebo + PEG + RBV | Cohort I - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort I - 3. Boceprevir + PEG + RBV - 44 Weeks | Cohort II - 1. Placebo + PEG + RBV | Cohort II - 2. Boceprevir + PEG + RBV - 24 Weeks (RGT) | Cohort II - 3. Boceprevir + PEG + RBV - 44 Weeks
Number analyzed (Participants) | 311 | 316 | 311 | 52 | 52 | 55
Participants
  Treatment week 4 (n=28, 18, 20, 2, 1, 0) | 27 | 16 | 18 | 2 | 1 | 0
  Treatment week 8 (n=56, 190, 182, 4, 18, 22) | 48 | 170 | 166 | 3 | 14 | 18
  Treatment week 12 (n=108, 237, 231, 10, 25, 33) | 90 | 205 | 204 | 7 | 19 | 26
  Treatment week 16 (n=138, 231, 237, 15, 26, 36) | 106 | 205 | 210 | 12 | 20 | 26
  Treatment week 20 (n=157, 231, 231, 15, 27, 32) | 118 | 201 | 208 | 12 | 21 | 26

ADVERSE EVENTS:
Groups:
- PEG + RBV: Cohort I (White participants) and Cohort II (Black participants) treated with PegIntron (PEG) 1.5 μg/kg + Ribavirin (RBV) (weight-based dosing [WBD]) for 4 weeks followed by placebo + PEG 1.5 μg/kg + RBV (WBD) for 44 weeks with 24 weeks post-treatment follow-up.
- BOCEPREVIR + PEG + RBV - 24 WEEKS: Cohort I (White participants) and Cohort II (Black participants) treated with PEG 1.5 μg/kg + RBV (WBD) for 4 weeks followed by boceprevir + PEG 1.5 μg/kg + RBV (WBD) for 24 weeks. Participants were offered a response guided therapy (RGT) at treatment week 28.
  * At the Treatment Week 28 visit, participants whose HCV-RNA was undetectable at Treatment Week 8 and at all subsequent assays (up to Treatment Week 24), will proceed to the 44-week follow-up.
  * At the Treatment Week 28 visit, participants with detectable HCV-RNA at Treatment Week 8 or at any subsequent assays will continue on therapy with placebo + PEG 1.5 μg/kg + RBV (WBD) for an additional 20 weeks, to complete a total of 48 weeks on treatment with 24 weeks post-treatment follow-up.
- BOCEPRIVIR + PEG + RBV - 44 WEEKS: Cohort I (White participants) and Cohort II (Black participants) treated with PEG 1.5 μg/kg + RBV (WBD) for 4 weeks followed by boceprevir + PEG 1.5 μg/kg + RBV (WBD) for 44 weeks with 24 weeks post-treatment follow-up.
Arm/Group | PEG + RBV | BOCEPREVIR + PEG + RBV - 24 WEEKS | BOCEPRIVIR + PEG + RBV - 44 WEEKS
Serious Adverse Events (participants affected / at risk) | 31/363 | 42/368 | 45/366
Other Adverse Events (participants affected / at risk) | 353/363 | 365/368 | 363/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG + RBV (N=363) | BOCEPREVIR + PEG + RBV - 24 WEEKS (N=368) | BOCEPRIVIR + PEG + RBV - 44 WEEKS (N=366)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 3 (5) | 4 (7)
APLASIA PURE RED CELL (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (3)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTROPHIC CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
DEAFNESS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
OPTIC NEUROPATHY (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
PAPILLOEDEMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COLONIC POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 2 (2)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 4 (4)
DEATH (General disorders) | 2 (2) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 1 (1) | 3 (3)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
CHOLELITHIASIS OBSTRUCTIVE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
SARCOIDOSIS (Immune system disorders) | 0 (0) | 0 (0) | 1 (2)
ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ATYPICAL MYCOBACTERIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
EPIGLOTTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
INFECTED BITES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INJECTION SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PERIRECTAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 3 (4) | 1 (1)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SCROTAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
TRACHEOBRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
MOTOR NEURONE DISEASE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASTICITY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
AFFECTIVE DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
ALCOHOL ABUSE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
BIPOLAR I DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
DRUG ABUSE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DRUG DEPENDENCE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
PERSONALITY DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
PSYCHIATRIC DECOMPENSATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0) | 4 (4)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
GLOMERULONEPHRITIS MINIMAL LESION (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
SCROTAL PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PLEURAL FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ALCOHOL USE (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
PHYSICAL ASSAULT (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
LARYNGEAL OPERATION (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
SKIN NEOPLASM EXCISION (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
ACCELERATED HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG + RBV (N=363) | BOCEPREVIR + PEG + RBV - 24 WEEKS (N=368) | BOCEPRIVIR + PEG + RBV - 44 WEEKS (N=366)
ANAEMIA (Blood and lymphatic system disorders) | 107 (188) | 182 (292) | 179 (352)
LEUKOPENIA (Blood and lymphatic system disorders) | 33 (81) | 31 (83) | 45 (126)
NEUTROPENIA (Blood and lymphatic system disorders) | 77 (208) | 91 (216) | 93 (257)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 7 (16) | 16 (50) | 19 (38)
DRY EYE (Eye disorders) | 16 (16) | 13 (13) | 22 (24)
VISION BLURRED (Eye disorders) | 14 (15) | 23 (25) | 22 (25)
ABDOMINAL PAIN (Gastrointestinal disorders) | 20 (30) | 25 (28) | 23 (28)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 32 (40) | 30 (41) | 44 (54)
CONSTIPATION (Gastrointestinal disorders) | 32 (34) | 22 (24) | 32 (34)
DIARRHOEA (Gastrointestinal disorders) | 79 (103) | 80 (104) | 100 (125)
DRY MOUTH (Gastrointestinal disorders) | 40 (45) | 39 (42) | 43 (51)
DYSPEPSIA (Gastrointestinal disorders) | 32 (39) | 29 (35) | 33 (40)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 8 (9) | 19 (22) | 20 (22)
NAUSEA (Gastrointestinal disorders) | 153 (199) | 175 (231) | 159 (212)
VOMITING (Gastrointestinal disorders) | 57 (70) | 75 (99) | 70 (90)
ASTHENIA (General disorders) | 70 (129) | 55 (86) | 70 (132)
CHILLS (General disorders) | 102 (114) | 134 (156) | 121 (139)
FATIGUE (General disorders) | 217 (279) | 196 (250) | 209 (290)
INFLUENZA LIKE ILLNESS (General disorders) | 93 (160) | 91 (113) | 83 (102)
INJECTION SITE ERYTHEMA (General disorders) | 47 (55) | 46 (48) | 37 (38)
INJECTION SITE REACTION (General disorders) | 44 (46) | 45 (46) | 39 (39)
IRRITABILITY (General disorders) | 86 (106) | 81 (104) | 83 (111)
PAIN (General disorders) | 34 (36) | 41 (43) | 37 (41)
PYREXIA (General disorders) | 120 (196) | 123 (180) | 117 (218)
SINUSITIS (Infections and infestations) | 15 (18) | 16 (20) | 19 (22)
WEIGHT DECREASED (Investigations) | 46 (54) | 43 (50) | 52 (64)
DECREASED APPETITE (Metabolism and nutrition disorders) | 90 (101) | 97 (107) | 89 (98)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 66 (84) | 69 (87) | 72 (103)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 40 (45) | 30 (33) | 40 (45)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 23 (25) | 15 (20) | 18 (20)
MYALGIA (Musculoskeletal and connective tissue disorders) | 94 (125) | 78 (98) | 92 (120)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 19 (21) | 11 (12) | 21 (24)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 27 (30) | 22 (23) | 18 (18)
DIZZINESS (Nervous system disorders) | 59 (74) | 80 (97) | 66 (70)
DYSGEUSIA (Nervous system disorders) | 64 (68) | 137 (143) | 156 (164)
HEADACHE (Nervous system disorders) | 153 (264) | 168 (233) | 167 (311)
MEMORY IMPAIRMENT (Nervous system disorders) | 21 (21) | 9 (9) | 24 (28)
PARAESTHESIA (Nervous system disorders) | 13 (32) | 10 (11) | 19 (23)
ANXIETY (Psychiatric disorders) | 42 (49) | 50 (57) | 48 (65)
DEPRESSION (Psychiatric disorders) | 78 (86) | 82 (103) | 69 (85)
INSOMNIA (Psychiatric disorders) | 118 (137) | 117 (145) | 122 (141)
MOOD SWINGS (Psychiatric disorders) | 6 (7) | 13 (17) | 19 (21)
COUGH (Respiratory, thoracic and mediastinal disorders) | 76 (87) | 56 (69) | 74 (100)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 59 (66) | 68 (87) | 84 (94)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 30 (33) | 42 (44) | 31 (39)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 19 (23) | 21 (21)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 22 (24) | 14 (18) | 33 (34)
ALOPECIA (Skin and subcutaneous tissue disorders) | 99 (105) | 75 (82) | 104 (109)
DRY SKIN (Skin and subcutaneous tissue disorders) | 66 (77) | 67 (72) | 86 (98)
PRURITUS (Skin and subcutaneous tissue disorders) | 98 (130) | 87 (101) | 94 (138)
RASH (Skin and subcutaneous tissue disorders) | 83 (124) | 93 (111) | 88 (119)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In this multicenter trial, initially, the investigator may only publish study results together with the other sites, unless specific written permission is obtained in advance from the sponsor.

The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a 45 day period from the time submitted to the sponsor for review.